CLINICAL TRIAL: NCT05686928
Title: A Multi-center, Prospective Pilot Study on Safety and Effectiveness of a Healing Ointment as a Post-surgical Care
Brief Title: Healing Ointment Usage Post-surgical Procedure
Acronym: Cetaphil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04.US.SL.017
Record Dates: First submitted 2022-11-07; First posted 2023-01-17 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Healing Ointment (Experimental): Petrolatum-based opaque ointment applied to surgical wound twice daily.
  Interventions: Drug: Cetaphil Healing Ointment

INTERVENTIONS:
Drug: Cetaphil Healing Ointment — Topical ointment application twice daily

SUMMARY:
To evaluate benefits of a Healing Ointment in skin improvement after dermatologic procedures

DETAILED DESCRIPTION:
This is an open-label, multi-center study to evaluate the safety and efficacy of a Healing Ointment in skin improvement after dermatologic procedures such as Mohs surgery, skin biopsy, excision on the head/neck or body.

The study is designed to enroll approximately 20 subjects, in which 10 subjects undergo dermatologic procedure on the head/neck and 10 subjects on the body.

Eligible subjects apply the test product twice daily after the procedure, followed by efficacy and tolerability assessments, standard photography, and self-assessment questionnaire at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject who undergo Mohs surgery, skin biopsy, excision on the head/neck or body
* Ability of giving consent for participation in the study
* Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments

Exclusion Criteria:

* History of allergy or hypersensitivity to cosmetic ingredients
* Pregnant, planning pregnancy during the course of the study or breastfeeding
* Subject with a history of keloids or hypertrophic scars
* Presence of tattoo and/or scar in the treatment area that in the investigator's opinion would interfere with study assessments
* Subjects with history of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis) at the discretion of the investigator
* Subjects with inability to comply with all study protocol restrictions and visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Farberg, MD, Principal Investigator — Derm Texas and Legacy Dermatology
Locations (2):
- United States (2):
  - Derm Texas, Dallas, Texas
  - Legacy Dermatology, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects met the inclusion and exclusion criteria, and were enrolled in the study.
Period: Overall Study
Arm/Group | Healing Ointment
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (21.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian Non-Hispanic | 10
  Race/Ethnicity: Hispanic | 5
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Erythema Assessment Using Clinical Grading Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Erythema assessment was graded clinically based on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.8 (0.68)
  Immediate post-procedure | 0.83 (0.65)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0.75 (0.64)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0.29 (0.45)

2. Primary Outcome: Objective Edema Assessment Using Clinical Grading Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Edema assessment was graded clinically based on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.03 (0.13)
  Immediate post-procedure | 0.5 (0.5)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0 (0)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0 (0)

3. Primary Outcome: Objective Overall Wound Appearance Assessment Using Clinical Grading Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Overall wound appearance was graded clinically based on a scale from 0 to 3 (0 = excellent, 1 = good, 2 = fair, 3 = poor).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.57 (0.88)
  Immediate post-procedure | 2.13 (0.48)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 1.36 (0.46)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0.54 (0.66)

4. Primary Outcome: Objective Scabbing/Crusting Assessment Using Clinical Grading Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Scabbing/crusting assessment was graded based on a scale from 0 to 4 (0 = none, 1 = slight, 2 = moderate, 3 = extensive, 4 = almost complete/complete).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.53 (0.83)
  Immediate post-procedure | 0 (0)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0.14 (0.31)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0 (0)

5. Primary Outcome: Subjective Burning Assessment Using an Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Burning assessment was graded by subjects based on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.2 (0.56)
  Immediate post-procedure | 0 (0)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0.04 (0.13)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0 (0)

6. Primary Outcome: Subjective Itching Assessment Using an Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Itching assessment was graded by subjects based on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.53 (0.74)
  Immediate post-procedure | 0.07 (0.26)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0.04 (0.13)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0 (0)

7. Primary Outcome: Subjective Pain Assessment Using an Analog Scale
Description: Summary of change in tolerability from baseline to day 28, at the surgical area after using the Healing Ointment daily. Lower scores reflect a better outcome. Pain assessment was graded by subjects based on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Immediately post-procedure (on the same day of the procedure), day 7/14, and day 28 from baseline
Population: Analysis population was based on Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Ointment
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.13 (0.52)
  Immediate post-procedure | 0 (0)
  Day 7/14: number analyzed (Participants) | 14
  Day 7/14 | 0 (0)
  Day 28: number analyzed (Participants) | 12
  Day 28 | 0 (0)

8. Secondary Outcome: Subject Satisfaction Using a Self-assessment Questionnaire
Description: Subjects are asked about their satisfaction with the treatment product and overall improvement at the treated area. Scale consists of 5 questions at every follow-up visit and subjects select level of satisfaction for each question from/to strongly agree, agree, neither, disagree, and strongly disagree. Upon study completion, subjects also provide their perception on recommendation, purchase intent, preference, and testimonial.
Time Frame: Day 7/14
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Ointment
Number analyzed (Participants) | 14
Participants
  Subjects reported the wound felt moisturized | 13
  Subjects reported the treatment product soothed the wound and surrounding skin | 13
  Subjects reported the treatment product improved the status of the wound | 13
  Subjects reported the treatment product did not irritate the wound area | 14

9. Secondary Outcome: Subject Satisfaction Using a Self-assessment Questionnaire
Description: as for outcome 8
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Ointment
Number analyzed (Participants) | 12
Participants
  Subjects reported the treatment product helped the wound heal effectively | 12
  Subjects reported the treatment product provided a protective layer for the wound | 12
  Subjects reported the treatment product kept the wound surface clean and moisturized | 11
  Subjects reported the treatment product did not feel greasy on their skin | 10

ADVERSE EVENTS:
Time Frame: 4 weeks (i.e., from the study start to the study completion).
Description: Throughout the course of the study, all adverse events were monitored and reported on an adverse event CRF/eCRF without omitting any requested and known information.
Arm/Group | Healing Ointment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT05686928/Prot_SAP_000.pdf